CLINICAL TRIAL: NCT01363011
Title: A Phase 3 Open-label Safety Study of Cobicistat-containing Highly Active Antiretroviral Regimens in HIV-1 Infected Patients With Mild to Moderate Renal Impairment
Brief Title: Cobicistat-containing Highly Active Antiretroviral Regimens in HIV-1 Infected Patients With Mild to Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0118
Record Dates: First submitted 2011-05-11; First posted 2011-06-01 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; Treatment Naive; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Cobicistat; Atazanavir Sulfate; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E/C/F/TDF (Cohort 1) (Experimental): Participants who have not received prior antiretroviral (ARV) treatment and who are virologically unsuppressed at baseline will initiate treatment with elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) single-tablet regimen (STR) for up to 96 weeks.
  Following Week 96, participants continued their treatment until all participants discontinued from the study or commercial approval of E/C/F/TDF was received in the applicable country.
  Interventions: Drug: E/C/F/TDF
- COBI+PI+2 NRTI (Cohort 2) (Experimental): Participants who have received prior ARV treatment and who are virologically suppressed at baseline will continue their treatment regimen, switching the regimen's pharmacoenhancer component from ritonavir to cobicistat (COBI), and continuing their existing protease inhibitor (PI; either atazanavir (ATV) or darunavir (DRV)) plus 2 nucleoside reverse transcriptase inhibitor (NRTI) regimen for up to 96 weeks.
  Following Week 96, participants continued their treatment until all participants discontinued from the study or commercial approval of cobicistat was received in the applicable country.
  Interventions: Drug: COBI; Drug: ATV; Drug: DRV; Drug: NRTI

INTERVENTIONS:
Drug: E/C/F/TDF — E/C/F/TDF (150/150/200/300 mg) STR administered orally once daily
  Other Names: Stribild®
  Arms: E/C/F/TDF (Cohort 1)
Drug: COBI — COBI 150 mg tablet administered with food orally once daily
  Other Names: Tybost®
  Arms: COBI+PI+2 NRTI (Cohort 2)
Drug: ATV — ATV 300 mg tablet administered orally once daily
  Other Names: Reyataz®
  Arms: COBI+PI+2 NRTI (Cohort 2)
Drug: DRV — DRV 800 mg tablet administered orally once daily
  Other Names: Prezista®
  Arms: COBI+PI+2 NRTI (Cohort 2)
Drug: NRTI — Participants will receive 2 investigator-selected NRTIs, which may include abacavir (ABC), lamivudine (3TC)/zidovudine (ZDV), didanosine (DDI), emtricitabine (FTC), ABC/3TC, 3TC, tenofovir disoproxil fumarate (TDF), or FTC/TDF, administered according to prescribing information.
  Arms: COBI+PI+2 NRTI (Cohort 2)

SUMMARY:
This study is to characterize the effect of cobicistat-based regimens on parameters of renal function in participants with HIV infection and who have mild to moderate renal impairment, and to assess the safety and tolerability of the regimens in order to generate appropriate dosing recommendations.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (treatment-naive)

* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* Screening genotype report must show sensitivity to FTC and TDF
* No prior use of any approved or investigational antiretroviral drug for any length of time

Cohort 2 (treatment-experienced, pharmacoenhancer switch)

* Subjects must be receiving ATV 300 mg/ritonavir (RTV) 100 mg plus 2 NRTIs OR DRV 800 mg/RTV 100 mg plus 2 NRTIs for at least 6 months prior to screening
* Plasma HIV-1 RNA concentrations at undetectable levels in the 6 months preceding the screening visit and have HIV-1 RNA < 50 copies/mL at screening
* Subjects experiencing intolerance to RTV (as determined by the investigator)

Both groups

* The ability to understand and sign a written informed consent form
* Normal ECG
* Mild to moderate renal function
* Stable renal function
* Hepatic transaminases (AST and ALT) ≤ 5 x the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin (subjects with documented Gilbert's Syndrome or hyperbilirubinemia due to atazanavir therapy may have total bilirubin up to 5 x ULN)
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Males and females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drug
* Age ≥ 18 years

Exclusion Criteria:

* New AIDS-defining condition diagnosed within the 30 days prior to screening
* Receiving drug treatment for hepatitis C, or anticipated to receive treatment for hepatitis C
* Subjects experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the investigator to potentially interfere with subject study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Receiving ongoing therapy with any of medications contraindicated for use with elvitegravir (EVG), COBI, FTC, TDF, ATV, DRV; or subjects with any known allergies to the excipients of E/C/F/TDF STR, COBI tablets, ATV capsules or DRV tablets or contraindicated for the 2 NRTIs as part of the PI/co regimen
* Participation in any other clinical trial without prior approval
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Szwarcberg, MD, Study Director — Gilead Sciences
Locations (51):
- United States (34):
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic, Little Rock, Arkansas
  - AHF Research Center, Beverly Hills, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, M.D., Inc., Los Angeles, California
  - Anthony Mills, MD, Inc., Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - East Bay AIDS Center, Oakland, California
  - University of California, Davis, Sacramento, California
  - Metropolis Medical, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine AIDS Program, New Haven, Connecticut
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Broward Health, Fort Lauderdale, Florida
  - Gary J. Richmond.M.D.,P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ValueHealthMD, LLC, Orlando, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University/ Mercer Medicine Clinical Research, Macon, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - The Research Institute, Springfield, Massachusetts
  - Central West Clinical Research, Inc., St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Chelsea Village Medical, New York, New York
  - Mount Sinai Downtown Comprehensive Health Program, New York, New York
  - AIDS Care, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Southwest Infectious Disease Clinical Research, Inc., Addison, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
- Australia (3):
  - Taylor Square Private Clinic, Darlinghurst
  - Infectious Diseases Unit - The Alfred Hospital, Melbourne
  - Holdsworth House Medical Practice, Sydney
- Austria (2):
  - Landeskrankenhaus Graz West, Graz
  - Otto Wagner Spital, Vienna
- Canada (2):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal
- Instituto Dominicano de Estudio Virologicos, Santo Domingo, Dominican Republic
- Center for HIV and Hepatogastroenterology, Düsseldorf, Germany
- Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Mexico
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan
  - HOPE Clinical Research, San Juan
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Barts & the London NHS Trust, London
  - Homerton University Hospital, London
  - Guy's King's and St. Thomas' School of Medicine, London
  - St Stephen's AIDS Trust, London

REFERENCES:
- [Result] Fisher M, McDonald C, Moyle G, Martorell C, Ramgopal M, Laplante F, Curley J, Graham H, Tran-Muchowski C, Liu Y, Rhee M, Szwarcberg J. Switching from ritonavir to cobicistat in HIV patients with renal impairment who are virologically suppressed on a protease inhibitor. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19824. doi: 10.7448/IAS.17.4.19824. eCollection 2014. PMID 25397568
- [Result] Post FA, Winston J, Andrade-Villanueva JF, Fisher M, Liu Y, Beraud C, Abram ME, Graham H, Rhee MS, Cheng AK, Szwarcberg J; Study 118 Team. Elvitegravir/cobicistat/emtricitabine/tenofovir DF in HIV-infected patients with mild-to-moderate renal impairment. J Acquir Immune Defic Syndr. 2015 Mar 1;68(3):310-3. doi: 10.1097/QAI.0000000000000476. PMID 25469527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 40 study sites in Australia, Europe, and North America. The first participant was screened on 13 May 2011. The last study visit occurred on 16 February 2015.
Pre-assignment Details: 177 participants were screened.
Groups:
- E/C/F/TDF (Cohort 1): Main Study: Participants who had not received prior antiretroviral (ARV) treatment and who were virologically unsuppressed at baseline initiated treatment with elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (Stribild®; E/C/F/TDF) (150/150/200/300 mg) single-tablet regimen (STR) once daily for up to 96 weeks.
  Extension Phase: Participants continued their treatment until all participants discontinued from the study or commercial approval of E/C/F/TDF was received in the applicable country.
- COBI+PI+2 NRTIs (Cohort 2): Main Study: Participants who had received prior ARV treatment and who were virologically suppressed at baseline switched their regimen's pharmacoenhancer component from ritonavir to cobicistat (Tybost®; COBI) 150 mg, while continuing the other components of their ARV regimen (atazanavir (ATV) 300 mg or darunavir (DRV) 800 mg plus 2 nucleoside reverse transcriptase inhibitors (NRTI)) for up to 96 weeks. These 2 NRTIs may have included abacavir (ABC), lamivudine (3TC)/zidovudine (ZDV), didanosine (DDI), emtricitabine (FTC), ABC/3TC, 3TC, tenofovir disoproxil fumarate (TDF), or emtricitabine/tenofovir disoproxil fumarate (Truvada®; FTC/TDF), administered according to prescribing information.
  Extension Phase: Participants continued their treatment until all participants discontinued from the study or commercial approval of cobicistat was received in the applicable country.
Period: Main Study
Arm/Group | E/C/F/TDF (Cohort 1) | COBI+PI+2 NRTIs (Cohort 2)
Started | 33 | 73
Completed | 29 | 64
Not Completed | 4 | 9
Not completed — Adverse Event | 2 | 3
Not completed — Investigator's Discretion | 1 | 1
Not completed — Withdrew Consent | 1 | 4
Not completed — Protocol Violation | 0 | 1
Period: Extension Phase
Arm/Group | E/C/F/TDF (Cohort 1) | COBI+PI+2 NRTIs (Cohort 2)
Started | 18 (11 participants who completed the main study did not enroll into the extension phase.) | 49 (15 participants who completed the main study did not enroll into the extension phase.)
Completed | 13 | 41
Not Completed | 5 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Investigator's Discretion | 2 | 2
Not completed — Withdrew Consent | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Rolled Over to Another Gilead Study | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug
Groups:
- E/C/F/TDF (Cohort 1): Main Study: Participants who had not received prior ARV treatment and who were virologically unsuppressed at baseline initiated treatment with E/C/F/TDF (150/150/200/300 mg) STR once daily for up to 96 weeks.
  Extension Phase: Participants continued their treatment until all participants discontinued from the study or commercial approval of E/C/F/TDF was received in the applicable country.
- COBI+PI+2 NRTIs (Cohort 2): Main Study: Participants who had received prior ARV treatment and who were virologically suppressed at baseline switched their regimen's pharmacoenhancer component from ritonavir to COBI 150 mg, while continuing the other components of their ARV regimen (ATV 300 mg or DRV 800 mg plus 2 NRTIs) for up to 96 weeks. These 2 NRTIs may have included ABC, 3TC/ZDV, DDI, FTC, ABC/3TC, 3TC, TDF, or FTC/TDF, administered according to prescribing information.
  Extension Phase: Participants continued their treatment until all participants discontinued from the study or commercial approval of cobicistat was received in the applicable country.
- Total: Total of all reporting groups
Arm/Group | E/C/F/TDF (Cohort 1) | COBI+PI+2 NRTIs (Cohort 2) | Total
Number analyzed (Participants) | 33 | 73 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.1) | 54 (9.5) | 53 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 27 | 60 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Black or African Heritage | 13 | 14 | 27
  White | 14 | 56 | 70
  Other | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 9 | 19 | 28
  Non-Hispanic/Latino | 24 | 54 | 78
Region of Enrollment [Number; unit: participants]
  United States | 19 | 33 | 52
  Mexico | 0 | 9 | 9
  Canada | 4 | 2 | 6
  Dominican Republic | 5 | 1 | 6
  Austria | 0 | 2 | 2
  Australia | 1 | 5 | 6
  Germany | 0 | 3 | 3
  United Kingdom | 4 | 18 | 22
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 28 | 37 | 65
  Symptomatic HIV Infection | 3 | 18 | 21
  AIDS | 2 | 18 | 20
Hepatitis B Virus (HBV) Surface Antigen Status [Number; unit: participants]
  Positive | 1 | 4 | 5
  Negative | 32 | 69 | 101
Hepatitis C Virus (HCV) Antibody Status [Number; unit: participants]
  Positive | 2 | 10 | 12
  Negative | 30 | 63 | 93
  Indeterminate | 1 | 0 | 1
HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 0 | 73 | 73
  ≥ 50 to < 1,000 copies/mL | 0 | 0 | 0
  ≥ 1,000 to ≤ 100,000 copies/mL | 24 | 0 | 24
  > 100,000 copies/mL | 9 | 0 | 9
CD4 Cell Count [Number; unit: participants]
  ≤ 50 cells/µL | 1 | 0 | 1
  51 to ≤ 200 cells/µL | 3 | 3 | 6
  201 to ≤ 350 cells/µL | 13 | 5 | 18
  351 to ≤ 500 cells/µL | 10 | 16 | 26
  > 500 cells/µL | 6 | 49 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) Using the Cockcroft-Gault (CG) Equation at Week 24 (Cohort 1)
Description: Change from baseline in eGFR-CG equation at Week 24 was analyzed in Cohort 1 (treatment-naive).
Time Frame: Baseline; Week 24
Population: Safety Analysis Set (treatment-naive only): participants in the treatment-naive group who were randomized and received at least one dose of study drug
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min
  Baseline (n = 33) | 72.9 [64.7 to 81.1]
  Change at Week 24 (n = 30) | -5.2 [-13.2 to 1.0]

2. Primary Outcome: Change From Baseline in eGFR-CG at Week 24 (Cohort 2)
Description: Change from baseline in eGFR-CG equation at Week 24 was analyzed in Cohort 2 (treatment-experienced).
Time Frame: Baseline; Week 24
Population: Safety Analysis Set (treatment-experienced only): participants in the treatment-experienced group who were randomized and received at least one dose of study drug
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min
  Baseline (n = 73) | 71.4 [61.9 to 80.7]
  Change at Week 24 (n = 67) | -3.7 [-7.4 to 2.0]

3. Secondary Outcome: Change From Baseline in eGFR-CG at Weeks 48 and 96 (Cohort 1)
Description: Change from baseline in eGFR-CG at Weeks 48 and 96 were analyzed in Cohort 1 (treatment-naive). This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min
  Change at Week 48 (n = 28) | -7.6 [-12.2 to -2.2]
  Change at Week 96 (n = 25) | -7.9 [-14.2 to -4.1]

4. Secondary Outcome: Change From Baseline in eGFR-CG at Weeks 48 and 96 (Cohort 2)
Description: Change from baseline in eGFR-CG at Weeks 48 and 96 were analyzed in Cohort 2 (treatment-experienced). This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set (treatment-experienced only) with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min
  Change at Week 48 (n = 63) | -3.8 [-9.0 to 0.8]
  Change at Week 96 (n = 50) | -5.0 [-13.0 to 0.1]

5. Secondary Outcome: Change From Baseline in eGFR-MDRD at Weeks 48 and 96 (Cohort 1)
Description: Change from baseline in eGFR-MDRD at Weeks 48 and 96 were analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Change at Week 48 (n = 28) | -12.1 [-17.6 to -6.5]
  Change at Week 96 (n = 25) | -12.9 [-17.7 to -5.4]

6. Secondary Outcome: Change From Baseline in eGFR-MDRD at Weeks 48 and 96 (Cohort 2)
Description: Change from baseline in eGFR-MDRD at Weeks 48 and 96 were analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Change at Week 48 (n = 63) | -3.9 [-8.1 to 1.4]
  Change at Week 96 (n = 50) | -2.8 [-13.7 to 2.2]

7. Secondary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation at Weeks 48 and 96 (Cohort 1)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (not adjusted for age, sex, and race) at Weeks 48 and 96 were analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Change at Week 48 (n = 28) | 1.9 [-7.1 to 6.9]
  Change at Week 96 (n = 25) | 12.4 [-0.6 to 20.4]

8. Secondary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation at Weeks 48 and 96 (Cohort 2)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (not adjusted for age, sex, and race) at Weeks 48 and 96 were analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Change at Week 48 (n = 63) | -4.7 [-12.0 to 4.3]
  Change at Week 96 (n = 50) | -2.4 [-7.3 to 9.4]

9. Primary Outcome: Change From Baseline in eGFR Using the Modification of Diet in Renal (MDRD) Equation at Week 24 (Cohort 1)
Description: Change from baseline in eGFR-MDRD equation at Week 24 was analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Baseline (n = 33) | 77.1 [64.3 to 87.2]
  Change at Week 24 (n = 30) | -7.4 [-16.3 to -1.2]

10. Primary Outcome: Change From Baseline in eGFR-MDRD at Week 24 (Cohort 2)
Description: Change from baseline in eGFR-MDRD equation at Week 24 was analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Baseline (n = 73) | 65.8 [56.2 to 75.2]
  Change at Week 24 (n = 67) | -3.4 [-7.5 to 1.9]

11. Primary Outcome: Change From Baseline in eGFR Using the Chronic Kidney Disease, Epidemiology Collaboration (CKD-EPI) Formula Based on Cystatin C Equation at Week 24 (Cohort 1)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (not adjusted for age, sex, and race) at Week 24 was analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Baseline (n = 33) | 77.6 [61.7 to 90.5]
  Change at Week 24 (n = 30) | 0.3 [-3.3 to 6.1]

12. Primary Outcome: Change From Baseline in eGFR-CKD-EPI Formula Based on Cystatin C Equation at Week 24 (Cohort 2)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (not adjusted for age, sex, and race) at Week 24 was analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Baseline (n = 73) | 78.6 [67.0 to 94.4]
  Change at Week 24 (n = 67) | -2.7 [-6.8 to 1.9]

13. Secondary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation (Adjusted) at Weeks 48 and 96 (Cohort 1)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (adjusted for age, sex, and race) at Weeks 48 and 96 were analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Change at Week 48 (n = 28) | 1.6 [-8.0 to 6.9]
  Change at Week 96 (n = 25) | 12.6 [-0.9 to 19.2]

14. Secondary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation (Adjusted) at Weeks 48 and 96 (Cohort 2)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (adjusted for age, sex, and race) at Weeks 48 and 96 were analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area. This outcome is to measure the long-term effect of COBI-containing regimens on renal parameters.
Time Frame: Baseline; Weeks 48 and 96
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Change at Week 48 (n = 63) | -4.7 [-11.7 to 3.9]
  Change at Week 96 (n = 50) | -2.8 [-7.4 to 8.9]

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 48 and 96 (Cohort 1)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Weeks 48 and 96 were analyzed in Cohort 1 (treatment-naive) using the FDA snapshot analysis algorithm.
Time Frame: Weeks 48 and 96
Population: Treatment-naive participants in the Full Analysis Set with available data was analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
percentage of participants
  Week 48 (n = 33) | 78.8
  Week 96 (n = 27) | 88.9

16. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 48 and 96 (Cohort 2)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Weeks 48 and 96 were analyzed in Cohort 2 (treatment-experienced) using the FDA snapshot analysis algorithm.
Time Frame: Weeks 48 and 96
Population: Treatment-experienced participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
percentage of participants
  Week 48 (n = 73) | 82.2
  Week 96 (n = 54) | 90.7

17. Secondary Outcome: Percentage of Participants Who Experienced Adverse Events (Cohort 1)
Description: Adverse events (AEs) occurring from baseline up to 30 days following the last dose of study drug were summarized for Cohort 1 (treatment-naive). A participant was counted once if they had a qualifying event.
Time Frame: Up to 147 weeks plus 30 days
Population: Safety Analysis Set (treatment-naive only)
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
percentage of participants
  Any AE | 100.0
  Drug-related AE | 48.5
  Grade 3 or higher AE | 21.2
  AE leading to drug discontinuation | 12.1
  Serious AE | 18.2
  AE of proximal renal tubulopathy | 0

18. Primary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation, Adjusted at Week 24 (Cohort 1)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (adjusted for age, sex, and race) at Week 24 was analyzed in Cohort 1 (treatment-naive). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-naive participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
mL/min/1.73 m^2
  Baseline (n = 33) | 76.9 [61.7 to 90.1]
  Change at Week 24 (n = 30) | 0.3 [-3.7 to 5.7]

19. Primary Outcome: Change From Baseline in eGFR-CKD-EPI Based on Cystatin C Equation, Adjusted at Week 24 (Cohort 2)
Description: Change from baseline in eGFR-CKD-EPI based on cystatin C equation (adjusted for age, sex, and race) at Week 24 was analyzed in Cohort 2 (treatment-experienced). The calculation was normalized to 1.73 m^2 body surface area.
Time Frame: Baseline; Week 24
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
mL/min/1.73 m^2
  Baseline (n = 73) | 78.2 [67.1 to 92.4]
  Change at Week 24 (n = 67) | -2.8 [-6.7 to 1.9]

20. Primary Outcome: Change From Baseline in Actual Glomerular Filtration Rate (aGFR) at Weeks 2, 4, and 24 (Cohort 1)
Description: Change from baseline in aGFR at Weeks 2, 4, and 24 was analyzed in Cohort 1 (treatment-naive). aGFR was calculated using iohexol plasma clearance.
Time Frame: Baseline; Weeks 2, 4, and 24
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) Substudy Analysis Set (treatment-naive only): participants in the treatment-naive group who were enrolled and received at least one dose of study drug and who had data for steady-state PK parameters at the relevant time points were analyzed.
Measure: Number; unit: mL/min
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
mL/min
  Baseline | 81.6
  Change at Week 2 | -12.1
  Change at Week 4 | -7.3
  Change at Week 24 | -3.3

21. Primary Outcome: Change From Baseline in aGFR at Weeks 2, 4, and 24 (Cohort 2)
Description: Change from baseline in aGFR at Weeks 2, 4, and 24 was analyzed in Cohort 2 (treatment-experienced). aGFR was calculated using iohexol plasma clearance.
Time Frame: Baseline; Weeks 2, 4, and 24
Population: PK/PD Substudy Analysis Set (treatment-experienced only): participants in the treatment-experienced group who were enrolled and received at least one dose of study drug and who had data for steady-state PK parameters at the relevant time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
mL/min
  Baseline | 82.5 [55.3 to 112.9]
  Change at Week 2 (n=13) | 1.6 [-12.3 to 9.2]
  Change at Week 4 (n=13) | 7.0 [-14.6 to 14.6]
  Change at Week 24 (n=11) | -4.1 [-13.5 to 13.2]

22. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 (Cohort 1)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed in Cohort 1 (treatment-naive) using the FDA snapshot analysis algorithm.
Time Frame: Week 24
Population: Full Analysis Set (treatment-naive only): participants in the treatment-naive group who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
percentage of participants | 84.8

23. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 (Cohort 2)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed in Cohort 2 (treatment-experienced) using the FDA snapshot analysis algorithm.
Time Frame: Week 24
Population: Full Analysis Set (treatment-experienced only): participants in the treatment-experienced group who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
percentage of participants | 90.4

24. Secondary Outcome: Percentage of Participants Who Experienced Adverse Events (Cohort 2)
Description: Adverse events (AEs) occurring from baseline up to 30 days following the last dose of study drug were summarized for Cohort 2 (treatment-experienced). A participant was counted once if they had a qualifying event.
Time Frame: Up to 166 weeks plus 30 days
Population: Safety Analysis Set (treatment-experienced only)
Measure: Number; unit: percentage of participants
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 73
percentage of participants
  Any AE | 93.2
  Drug-related AE | 27.4
  Grade 3 or higher AE | 28.8
  AE leading to drug discontinuation | 11.0
  Serious AE | 15.1
  AE of proximal renal tubulopathy | 0

25. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities (Cohort 1)
Description: Laboratory abnormalities were summarized for Cohort 1 (treatment-naive) and were defined as values that increased at least one toxicity grade from baseline at any time postbaseline up to and including the date of last dose of study drug plus 30 days. A participant was counted once if they had a qualifying event.
Time Frame: Up to 147 weeks plus 30 days
Population: Safety Analysis Set (treatment-naive only)
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 33
percentage of participants
  Any laboratory abnormality | 100.0
  Grade 3 or 4 laboratory abnormality | 39.4

26. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities (Cohort 2)
Description: Laboratory abnormalities were summarized for Cohort 2 (treatment-experienced) and were defined as values that increased at least one toxicity grade from baseline at any time postbaseline up to and including the date of last dose of study drug plus 30 days. A participant was counted once if they had a qualifying event.
Time Frame: Up to 166 weeks plus 30 days
Population: Treatment-experienced participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 72
percentage of participants
  Any laboratory abnormality | 100.00
  Grade 3 or 4 laboratory abnormality | 50.0

27. Secondary Outcome: Plasma Pharmacokinetics of COBI: AUCtau (Cohort 1)
Description: AUCtau was analyzed for Cohort 1 (treatment-naive) and was defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
Time Frame: Blood samples were collected at 0 (predose), 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 8.0, 12.0, and 24.0 hours postdose at baseline and Weeks 2, 4, and 24.
Population: PK/PD Substudy Analysis Set (treatment-naive only)
Measure: Number; unit: h*ng/mL
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
h*ng/mL
  Week 2 | 16554.7
  Week 4 | 12704.1
  Week 24 | 9799.7

28. Secondary Outcome: Plasma Pharmacokinetics of COBI: AUCtau (Cohort 2)
Description: AUCtau was analyzed for Cohort 2 (treatment-experienced) and was defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
Time Frame: as for outcome 27
Population: Participants in the PK/PD Substudy Analysis Set (treatment-experienced only) with available postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
h*ng/mL
  Week 2 (n = 13) | 12458.0 (6179.06)
  Week 4 (n = 13) | 11165.3 (4185.86)
  Week 24 (n = 11) | 13980.5 (8029.03)

29. Secondary Outcome: Plasma Pharmacokinetics of COBI: Cmax (Cohort 1)
Description: Cmax was analyzed for Cohort 1 (treatment-naive) and was defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 27
Population: PK/PD Substudy Analysis Set (treatment-naive only)
Measure: Number; unit: ng/mL
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
ng/mL
  Week 2 | 1734.6
  Week 4 | 1522.9
  Week 24 | 1266.4

30. Secondary Outcome: Plasma Pharmacokinetics of COBI: Cmax (Cohort 2)
Description: Cmax was analyzed for Cohort 2 (treatment-experienced) and was defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 27
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
ng/mL
  Week 2 (n = 13) | 1366.7 (508.32)
  Week 4 (n = 13) | 1297.7 (424.06)
  Week 24 (n = 11) | 1568.6 (618.84)

31. Secondary Outcome: Plasma Pharmacokinetics of COBI: Ctau (Cohort 1)
Description: Ctau was analyzed for Cohort 1 (treatment-naive) and was defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 27
Population: PK/PD Substudy Analysis Set (treatment-naive only)
Measure: Number; unit: ng/mL
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
ng/mL
  Week 2 | 150.5
  Week 4 | 37.3
  Week 24 | 24.2

32. Secondary Outcome: Plasma Pharmacokinetics of COBI: Ctau (Cohort 2)
Description: Ctau was analyzed for Cohort 2 (treatment-experienced) and was defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 27
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
ng/mL
  Week 2 (n = 13) | 79.9 (79.01)
  Week 4 (n = 13) | 71.3 (61.27)
  Week 24 (n = 11) | 139.8 (238.84)

33. Secondary Outcome: Plasma Pharmacokinetics of COBI: Tmax (Cohort 1)
Description: Tmax was analyzed for Cohort 1 (treatment-naive) and was defined as the time of Cmax.
Time Frame: as for outcome 27
Population: PK/PD Substudy Analysis Set (treatment-naive only)
Measure: Number; unit: hours
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
hours
  Week 2 | 4.00
  Week 4 | 2.00
  Week 24 | 4.00

34. Secondary Outcome: Plasma Pharmacokinetics of COBI: Tmax (Cohort 2)
Description: Tmax was analyzed for Cohort 2 (treatment-experienced) and was defined as the time of Cmax.
Time Frame: as for outcome 27
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
hours
  Week 2 (n = 13) | 3.92 [3.00 to 4.92]
  Week 4 (n = 13) | 4.92 [3.02 to 5.00]
  Week 24 (n = 11) | 3.00 [2.00 to 4.05]

35. Secondary Outcome: Plasma Pharmacokinetics of COBI: t1/2 (Cohort 1)
Description: t1/2 was analyzed for Cohort 1 (treatment-naive) and was defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 27
Population: PK/PD Substudy Analysis Set (treatment-naive only)
Measure: Number; unit: hours
Arm/Group | E/C/F/TDF (Cohort 1)
Number analyzed (Participants) | 1
hours
  Week 2 | 6.14
  Week 4 | 3.57
  Week 24 | 3.63

36. Secondary Outcome: Plasma Pharmacokinetics of COBI: t1/2 (Cohort 2)
Description: t1/2 was analyzed for Cohort 2 (treatment-experienced) and was defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 27
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | COBI+PI+2 NRTIs (Cohort 2)
Number analyzed (Participants) | 14
hours
  Week 2 (n = 13) | 4.37 [3.63 to 4.91]
  Week 4 (n = 12) | 3.98 [3.53 to 4.34]
  Week 24 (n = 10) | 3.77 [3.46 to 3.95]

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average: Cohort 1 = 93.7 weeks; Cohort 2 = 101.2 weeks) plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least one dose of study drug
Groups:
- COBI+PI+2 NRTIs (Cohort 2): Main Study: Participants who had received prior ARV treatment and who were virologically suppressed at baseline switched their regimen's pharmacoenhancer component from ritonavir to COBI 150 mg, while continuing the other components of their ARV regimen (ATV 300 mg or DRV 800 mg plus 2 NRTI) for up to 96 weeks. These 2 NRTIs may have included ABC, 3TC/ZDV, DDI, FTC, ABC/3TC, 3TC, TDF, or FTC/TDF, administered according to prescribing information.
  Extension Phase: Participants continued their treatment until all participants discontinued from the study or commercial approval of cobicistat was received in the applicable country.
Arm/Group | E/C/F/TDF (Cohort 1) | COBI+PI+2 NRTIs (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 6/33 | 11/73
Other Adverse Events (participants affected / at risk) | 31/33 | 66/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TDF (Cohort 1) (N=33) | COBI+PI+2 NRTIs (Cohort 2) (N=73)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TDF (Cohort 1) (N=33) | COBI+PI+2 NRTIs (Cohort 2) (N=73)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Vision blurred (Eye disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 12 | 10
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 9
Proctalgia (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4
Fatigue (General disorders) | 3 | 5
Oedema peripheral (General disorders) | 3 | 5
Pain (General disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 8
Acute sinusitis (Infections and infestations) | 1 | 4
Bronchitis (Infections and infestations) | 3 | 10
Chikungunya virus infection (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 4
Folliculitis (Infections and infestations) | 2 | 5
Gastroenteritis (Infections and infestations) | 2 | 2
Herpes simplex (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 4 | 8
Lower respiratory tract infection (Infections and infestations) | 1 | 5
Nasopharyngitis (Infections and infestations) | 6 | 14
Oral candidiasis (Infections and infestations) | 3 | 1
Pyuria (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 2 | 4
Sinusitis (Infections and infestations) | 4 | 7
Syphilis (Infections and infestations) | 4 | 1
Tinea cruris (Infections and infestations) | 2 | 0
Tinea pedis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 15
Urethritis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 5 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 2
Glomerular filtration rate decreased (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Dizziness (Nervous system disorders) | 3 | 7
Headache (Nervous system disorders) | 6 | 10
Abnormal dreams (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 7 | 6
Haematuria (Renal and urinary disorders) | 1 | 6
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal cyst (Renal and urinary disorders) | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 5
Hypertension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years